CLINICAL TRIAL: NCT06001099
Title: Gynecological Malignancies Earlystage Detection by Multi-omics Based Liquid Biopsy in Peripheral Blood: a Prospective, Extended Validation Study
Brief Title: PERformance of Multi-Cancer Early-detectIon Based on Various Biomarkers in fEmale Cancers, PERCEIVE-II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhong Zheng MD, Department of Gynecological Oncology, Fudan University Shanghai Cancer Center, Fudan University
Other Study IDs: RSCD2021002
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Gynecologic Cancer
Keywords: gynecologic cancer; early detection; liquid biopsy; cell-free DNA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, white blood cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer arm: Participants with new diagnosis of gynecologic cancers, from whom blood samples will be collected
- Healthy arm: Participants without a known cancer or certain benign disease, from whom blood samples will be collected

SUMMARY:
This study is a prospective study aimed to validate the performance of combined multi-omitcs assays for early detection of gynecologic cancers. Biomarkers of cfDNA methylation, ctDNA mutation and blood miRNA markers will be evaluated. The study will enroll approximately 2935 female participants, including participants with gynecologic cancers patients and healthy participants.

ELIGIBILITY:
Inclusion Criteria for Cancer Arm Participants:

* Age 18 years or older
* Able to provide a written informed consent
* Confirmed diagnosis or highly suspicious cases of gynecologic malignancies within 42 days prior to blood collection
* No prior or ongoing anti-cancer therapy (local or systematic) prior to study blood draw

Exclusion Criteria for Cancer Arm Participants:

* Pregnancy or lactating women
* Recipients of organ transplant or prior non-autologous (allogeneic) bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 7 days prior to study blood draw
* Recipients of any anti-cancer therapy within 30 days prior to study blood draw, due to diseases other than cancer.
* previous history of malignant tumor;
* precancerous lesions or benign diseases confirmed by biopsy or surgical specimen;
* unknown or insufficient to determine the nature of the lesion by histopathological reports;

Inclusion Criteria for healthy control Arm Participants:

* Able to provide a written informed consent.
* Able to provide sufficient and qualified blood samples for study tests.
* No cancer related symptoms within 30 days prior to study screening.
* Cancer history with curative treatment completed over 3 years without recurrence prior to study enrollment.

Exclusion Criteria for healthy control Arm Participants:

* Insufficient qualified blood sample for study test.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 30 days prior to study blood draw.
* Recipient of anti-infectious therapy within 14 days prior to study blood draw.
* Have received or are undergoing curative cancer treatment within three years prior to study screening.
* With autoimmune or other diseases with severe comorbidities.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from the participating medical center and assigned into two arms, including participants with new diagnosis of gynecologic malignancies and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 2935 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To validate the sensitivity, specificity and accuracy of tissue traceability of an early detection model based on combined cfDNA methylation and serum tumor markers in patients with gynecological malignancies | 24 months

SECONDARY OUTCOMES:
To verify the sensitivity, specificity and tissue traceability accuracy of cfDNA methylation as an early detection model for gynecological malignancies. | 24months
To verify the sensitivity and specificity of serum tumor markers alone as an early detection model for gynecological malignant tumors | 24months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, MD.&PHD, Principal Investigator — Department of Gynecological Oncology, Fudan University Shanghai Cancer Center
Locations (1):
- Fudan university shanghai cancer center, Deparment of gynecologic oncology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No